CLINICAL TRIAL: NCT00028691
Title: Chlorambucil Versus 2x2 Gy Involved Field Radiotherapy in Stage III/IV Previously Untreated Follicular Lymphoma Patients. A Prospective, Randomized Phase III Clinical Trial
Brief Title: Chlorambucil Compared With Radiation Therapy in Treating Patients With Previously Untreated Stage III or Stage IV Follicular Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Commissie Voor Klinisch Toegepast Onderzoek (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069120; CKVO-2001-01; HOVON-47NHL; EU-20131; HOVON-CKTO-2001-01; EORTC-20013
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2002-01

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Chlorambucil; Radiotherapy

INTERVENTIONS:
Drug: chlorambucil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. It is not yet known if chlorambucil is more effective than radiation therapy in treating follicular lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of chlorambucil with that of radiation therapy in treating patients who have stage III or stage IV follicular lymphoma that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of chlorambucil vs involved-field radiotherapy on progression-free survival of patients with previously untreated stage III or IV follicular lymphoma.
* Compare the complete and partial remission rates and overall survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral chlorambucil on days 1-5. Treatment repeats every 4 weeks for 6-8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients undergo radiotherapy on days 1 and 3 (and days 15 and 17 for split course).

Quality of life is assessed at baseline, prior to course 3, 6, and 8 (arm I), and then at 4-6 weeks after study.

Patients are followed at 4-6 weeks, 3-4 months (arm I), 3 months and 6 months (arm II), 11, 12, 15, 18, and 21 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 444 patients (222 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of follicular lymphoma

  * Stage III or IV disease
  * Grades I, II, or III
  * Previously untreated disease
* Nodal and extranodal sites
* Bidimensionally measurable disease by physical examination or diagnostic imaging
* No CNS or orbital non-Hodgkin's lymphoma localization

PATIENT CHARACTERISTICS:

Age:

* 18 and over (for patients at EORTC centers)
* 65 and over (for patients at HOVON centers)

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 6.0 g/dL

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No severe cardiac disease that would preclude study treatment

Pulmonary:

* No severe pulmonary disease that would preclude study treatment

Other:

* HIV negative
* No severe neurologic, psychiatric, or metabolic disease that would preclude study treatment
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No concurrent systemic corticosteroids, including dexamethasone for nausea and vomiting palliation (inhalation and topical corticosteroids allowed)

Radiotherapy:

* No concurrent elective radiotherapy to an adjacent negative lymph node

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Rick L. M. Haas, MD — The Netherlands Cancer Institute; T. Girinsky, MD — Gustave Roussy, Cancer Campus, Grand Paris
Locations (11):
- Algemeen Ziekenhuis Middelheim, Antwerp, Belgium
- Institut Gustave Roussy, Villejuif, France
- Netherlands (9):
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Akademisch Medisch Centrum, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Academisch Ziekenhuis Groningen, Groningen
  - Maastro Clinic, Heerlen
  - Leiden University Medical Center, Leiden
  - Radiotherapeutisch Instituut Limburg-Maastricht, Maastricht
  - Daniel Den Hoed Cancer Center at Erasmus University Medical Center, Rotterdam

REFERENCES:
- [Result] Haas RL, Girinsky T. HOVON 47/EORTC 20013: chlorambucil vs 2x2 Gy involved field radiotherapy in stage III/IV previously untreated follicular lymphoma patients. Ann Hematol. 2003 Jul;82(7):458-62. doi: 10.1007/s00277-003-0655-8. Epub 2003 May 20. No abstract available. PMID 12756499